CLINICAL TRIAL: NCT00461591
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Phase 3 Trial of Single Dose Intravesical Apaziquone (EOquin®) as a Surgical Adjuvant Instilled in the Early Postoperative Period in Patients Undergoing Transurethral Resection for Noninvasive Bladder Cancer (Protocol SPI-611)
Brief Title: Single Dose Intravesical Apaziquone Postoperative in Patients Undergoing TURBT for Noninvasive Bladder Cancer (SPI-611)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-611
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Bladder Cancer
Keywords: Noninvasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apaziquone (Experimental): TURBT + a single intravesical dose of Apaziquone 4mg in 40ml instilled into the bladder post-TURBT
  Interventions: Drug: Apaziquone; Procedure: TURBT
- Placebo (Placebo Comparator): TURBT + a single intravesical dose of placebo instilled into the bladder post-TURBT
  Interventions: Drug: Placebo; Procedure: TURBT

INTERVENTIONS:
Drug: Apaziquone — A single intravesical dose of Apaziquone 4mg in 40ml instilled into the bladder post-TURBT
  Other Names: EOquin®, Qapzola
  Arms: Apaziquone
Drug: Placebo — A single intravesical dose of placebo instilled into the bladder post-TURBT
  Arms: Placebo
Procedure: TURBT — TransUrethral Resection of the Bladder Tumor

SUMMARY:
The purpose of this study was to evaluate the 2-Year Recurrence Rate of bladder cancer in randomized patients with tumor histology Ta, G1-G2 who received TransUrethral Resection of Bladder Tumor (TURBT) plus apaziquone versus those who received TURBT plus placebo.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled study. Within 14 days of Screening, eligible patients underwent a TURBT during Visit 1 (Day 0) following which they were immediately randomized in a 1:1 ratio to receive either placebo or 4 mg apaziquone, instilled in a volume of 40 mL into the bladder within 6 hours from the end of the TURBT procedure. After a 60-minute retention period, study drug was drained from the bladder.

A postoperative follow-up examination and review of the local pathology report were performed at Visit 2, which occurred 21 days (±10 days) after the TURBT (Week 3).

* If the histology of the patient's tumor was confirmed as Ta, G1-G2 (ie, low grade according to World Health Organization [WHO]/International Society of Urologic Pathology [ISUP] classification), no further treatment was given and the patient was observed cystoscopically every 3 months through Year 2 for tumor recurrence (Visit 3 through Visit 10).
* If the histology of the patient's tumor was other than Ta, G1 or G2 (low grade [WHO/ISUP classification]), further treatment was given in accordance with current treatment guidelines, and the patient was followed up cystoscopically every 3 months through Year 2 for tumor recurrence (Visit 3 through Visit 10).

All patients were to be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria: (All questions must be answered YES)

* Has the patient given written informed consent?
* Is the patient at least 18 years old?
* Does the patient have transitional cell carcinoma of the bladder with clinically apparent stage Ta, grade G1-G2?
* If the patient is a female of childbearing potential, is she using an acceptable/effective method of contraception?
* If the patient is a female of childbearing potential, has she had a negative serum pregnancy test within the past 14 days?
* Is the patient willing and able to abide by the protocol?

Exclusion Criteria: (All questions must be answered NO)

* Does the patient have more than 4 bladder tumors?
* Does any single bladder tumor exceed 3.5 cm in diameter?
* Does the patient have a single, primary (no previous diagnosis of TCC) bladder tumor <0.5 cm?
* Has the patient ever received Apaziquone?
* Does the patient have, or has the patient ever had, any bladder tumor known to be other than stage Ta or grade G1 or G2 (low grade [WHO/ISUP classification])?
* Does the patient have, or has the patient ever had any bladder tumor with histology other than transitional cell carcinoma?
* Does the patient have, or has the patient ever had, carcinoma in situ (CIS)?
* Does the patient have an active urinary tract infection?
* Does the patient have a bleeding disorder or a screening platelet count < 100 x 10^9/L?
* Does the patient have any unstable medical condition that would make it unsafe for him/her to undergo TURBT under general or spinal anesthesia?
* Does the patient have a screening hemoglobin < 10 mg/dL, a screening absolute neutrophil count < 1.5 x 10^9/L or a screening creatinine > 2 mg/dL?
* Does the patient have a known immunodeficiency disorder?
* Has the patient received any investigational treatment within the past 30 days?
* Is the patient breast feeding?
* Does the patient have a history of interstitial cystitis?
* Does the patient have a history of allergy to red color food dye?
* Has the patient had transitional cell carcinoma of the bladder within the past 4 months?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (73):
- United States (73):
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - BCG Oncology, Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - Urology Associates Medical Group, Burbank, California
  - Urology Associates of Central CA, Fresno, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cancer Research Dept/St. Joseph Hospital, Orange, California
  - San Bernardino Urologic Association, San Bernardino, California
  - VA Medical Center, San Francisco, California
  - The Urology Center of Colorado, Denver, Colorado
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - Urologic Surgeons of Washington, Washington D.C., District of Columbia
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Urology Consultants, Longwood, Florida
  - University of Miami, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Florida Urology Specialists, Sarasota, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Gainesville Urology, PC, Gainesville, Georgia
  - Urological Professional Association, Macon, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, P.A., Meridian, Idaho
  - University of Chicago, Chicago, Illinois
  - Urology Associates, SC, Mattoon, Illinois
  - Speciality Care Research, Peoria, Illinois
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Kansas City Urology Care, P.A., Overland Park, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - Anne Arundel Urology, Annapolis, Maryland
  - Myron Murdock, MD, LLC, Greenbelt, Maryland
  - MMPC Urology, Grand Rapids, Michigan
  - Lakeside Urology, PC, Saint Joseph, Michigan
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Five Valleys Urology, Missoula, Montana
  - Coastal Urological Associates, PA, Brick, New Jersey
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Delaware Valley Urology, LLC-Marlton, Marlton, New Jersey
  - Deleware Valley Urology, LLC-Washington Township, Sewell, New Jersey
  - Delaware Valley Urology, LLC - Voorhees, Voorhees Township, New Jersey
  - Delaware Valley Urology, LLC-Westampton, Woodlane, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - Capital Region Urological Surgeons, Albany, New York
  - The Urological Institute of NE NY, Albany, New York
  - Adult and Pediatric Urology, Carmel, New York
  - Accumed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island, P.C., Garden City, New York
  - Hudson Valley Urology, PC, Kingston, New York
  - University Urology Associates, New York, New York
  - CNY Urology, PC, Oneida, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Urology Associates of Rochester, LLC, Rochester, New York
  - Center for Urologic Research of WNY, LLC, Williamsville, New York
  - TriState Urologic Services PSC, Inc., Cincinnati, Ohio
  - Columbus Urology Research, LLC, Columbus, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Urologic Consultants of South Eastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Triangle Urology Group, Pittsburgh, Pennsylvania
  - Susquehenna Urology, Williamsport, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Corpus Christi Urology Group LLC, Corpus Christi, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Mary Washington Hospital and Urology Associates of Fredericksburg, Fredericksburg, Virginia
  - Urology of Virginia, PC, Norfolk, Virginia
  - Urology of Virginia, PC, Virginia Beach, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - Seattle Urological Associates, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Apaziquone: Apaziquone: TURBT + a single intravesical dose of Apaziquone 4mg in 40ml instilled into the bladder post-TURBT
- Placebo: Placebo: TURBT + a single intravesical dose of placebo instilled into the bladder post-TURBT
Period: Overall Study
Arm/Group | Apaziquone | Placebo
Started | 406 | 396
Completed | 317 | 311
Not Completed | 89 | 85

BASELINE CHARACTERISTICS:
Population: Safety/ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Apaziquone | Placebo | Total
Number analyzed (Participants) | 406 | 396 | 802
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.92) | 68.2 (10.72) | 67.8 (10.82)
Age, Customized [Count of Participants; unit: Participants]
  Age: <65 | 159 | 146 | 305
  Age: 65-75 | 140 | 139 | 279
  Age: >75 | 107 | 111 | 218
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 102 | 210
  Male | 298 | 294 | 592
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 393 | 379 | 772
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 392 | 383 | 775
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 381 | 375 | 756
  Poland | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate at 2 Years
Description: The percentage of participants with histologically confirmed recurrence of the bladder tumor at any time after randomization and on or before year 2.
Time Frame: 2 years
Population: Target Ta, G1-G2 Population: patients who had 4 or fewer tumors that were ≤ 3.5 cm each at the time of randomization and who had subsequent histological confirmation from the central pathology lab that the tumors resected at the time of randomization were Ta, Grade 1 or 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
Participants
  Recurrence | 112 | 121
  Non-Recurrence | 183 | 150
Statistical Analysis 1: Comparison: Apaziquone vs Placebo; Test type: Superiority; p = 0.1068, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.54 to 1.06]

2. Secondary Outcome: Time to Recurrence
Description: The number of months from randomization to histologically confirmed recurrence of the patient's bladder tumor.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
months | 18.3 (0.47) | 16.7 (0.55)
Statistical Analysis 1: Comparison: Apaziquone vs Placebo; Test type: Superiority; p = 0.0412, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.59 to 0.99]

3. Secondary Outcome: Progression Rate at 2 Years
Description: The percentage of participants that progress to either a higher stage or grade from the histologically confirmed stage and grade at time of randomization.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
Participants
  Progression | 30 | 39
  Non-Progression | 265 | 232

4. Secondary Outcome: Time to Progression
Description: The number of months from randomization to progression to either a higher stage or grade of the patient's bladder tumor.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
months | 22.9 (0.26) | 22.0 (0.34)

5. Secondary Outcome: Number of Recurrences Per Patient
Description: The number of histologically confirmed recurrences during the course of the study.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: times
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
times | 0.6 (1.03) | 0.9 (1.21)

6. Secondary Outcome: Disease Free Interval
Description: The number of months from randomization to histologically confirmed progression of the patient's bladder tumor or death from any cause
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
months | 22.9 (0.26) | 22.0 (0.34)

7. Secondary Outcome: Disease Free Survival
Description: The number of months from randomization to histologically confirmed recurrence of the patient's bladder tumor or death from any cause
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
months | 18.0 (0.48) | 16.4 (0.55)

8. Secondary Outcome: Overall Survival
Description: The number of months from randomization to death from any cause.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 295 | 271
months | 20.3 (0.13) | 23.7 (0.14)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (ie, AEs that occurred or worsened following the TURBT procedure) were recorded from the time of randomization to Month 6; after Month 6 until Month 24 (end of study), only genitourinary AEs and Serious AEs (SAEs) were recorded.
Arm/Group | Apaziquone | Placebo
All-Cause Mortality (participants affected / at risk) | 11/406 | 13/396
Serious Adverse Events (participants affected / at risk) | 93/406 | 98/396
Other Adverse Events (participants affected / at risk) | 312/406 | 285/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apaziquone (N=406) | Placebo (N=396)
Hematuria (Renal and urinary disorders) | 6 | 8
Atrial Fibrillation (Cardiac disorders) | 6 | 0
Pneumonia (Infections and infestations) | 5 | 7
Cardiac Failure Congestive (Cardiac disorders) | 5 | 6
Chest Pain (General disorders) | 5 | 4
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Cellulitis (Infections and infestations) | 5 | 3
Hip Arthroplasty (Surgical and medical procedures) | 4 | 2
Coronary Artery Disease (Cardiac disorders) | 3 | 6
Knee Arthroplasty (Surgical and medical procedures) | 3 | 4
Myocardial Infarction (Cardiac disorders) | 3 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Syncope (Nervous system disorders) | 3 | 2
Urinary Bladder Hemorrhage (Renal and urinary disorders) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 5
Sepsis (Infections and infestations) | 2 | 3
Renal Failure Acute (Renal and urinary disorders) | 2 | 2
Acute Myocardial Infarction (Cardiac disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Transient Ischemic Attack (Nervous system disorders) | 2 | 1
Acute Coronary Syndrome (Cardiac disorders) | 2 | 0
Death (General disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Calculus ureteric (Renal and urinary disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 2
Anemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Ischemic ulcer (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Post procedural hematuria (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery disease (Nervous system disorders) | 1 | 0
Cerebrospinal fluid retention (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Angioplasty (Surgical and medical procedures) | 1 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Carotid endarterectomy (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Mitral valve replacement (Surgical and medical procedures) | 1 | 0
Penile prosthesis insertion (Surgical and medical procedures) | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 1 | 0
Labile hypertension (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Colitis ischemic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral hemorrhage (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder neoplasm surgery (Surgical and medical procedures) | 0 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 1
Radical prostatectomy (Surgical and medical procedures) | 0 | 1
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apaziquone (N=406) | Placebo (N=396)
Urinary tract infection (Infections and infestations) | 70 | 58
Procedural pain (Injury, poisoning and procedural complications) | 31 | 27
Bladder pain (Renal and urinary disorders) | 22 | 18
Bladder spasm (Renal and urinary disorders) | 29 | 23
Dysuria (Renal and urinary disorders) | 74 | 67
Haematuria (Renal and urinary disorders) | 38 | 57
Micturition urgency (Renal and urinary disorders) | 31 | 37
Pollakiuria (Renal and urinary disorders) | 39 | 46
Urinary retention (Renal and urinary disorders) | 17 | 30
Nausea (Gastrointestinal disorders) | 16 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication is the multi-center publication of Study results from all study sites. Other than the multi-center publication, site may publish an independent publication of data generated by site subject to Sponsor review rights (e.g., review for intellectual property, confidentiality).